CLINICAL TRIAL: NCT06165185
Title: Water and Coffee Intervention in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2010_740
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Excess Intake of Macronutrients; Excess Intake of Micronutrients; Vasopressin Low
Keywords: copeptin, water, coffee
MeSH Terms: conditions — Diabetes Insipidus | interventions — Water; Coffee

STUDY DESIGN:
Intervention Model Description: All subjects will be exposed to three different intervention procedures; water and coffee loads (acutely and chronically), or no change from usual fluid intake (as a time-control), respectively in randomized order. The daily intake of coffee or water will amount to 3 L of water and 1 L of coffee, respectively for one week each. 3 weeks of wash-out between each intervention week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water (Experimental): At intervention day 1, during a maximum time period of 20 minutes, subjects will ingest 1 L of water (still bottled water) to map the acute water effect on the vasopressin marker copeptin (repeated blood sampling every 30 minutes for 4 hours). Day 1 then continues with the rest of the daily intake, i.e., 2 L of extra water (i.e. in addition to each subject's habitual food and fluid intake).
  Intervention day 2-7: 3 L extra water per day in addition to each subject's habitual food and fluid intake.
  Interventions: Other: Water
- Coffee (Experimental): At intervention day 1, during a maximum time period of 20 minutes, subjects will ingest 4 dL of coffee to map the acute coffee effect on the vasopressin marker copeptin (repeated blood sampling every 30 minutes for 4 hours). Day 1 then continues with the rest of the daily intake, i.e., 6dL of extra coffee (i.e. in addition to each subject's habitual food and fluid intake).
  Intervention day 2-7: 1 L extra coffee per day in addition to each subject's habitual food and fluid intake.
  Interventions: Other: Coffee
- Control (Experimental): At intervention day 1, during a maximum time period of 20 minutes, subjects will ingest just 10 ml of water to map the acute effect on the vasopressin marker copeptin (repeated blood sampling every 30 minutes for 4 hours). Day 1 then continues with each subject's habitual food and fluid intake.
  Intervention day 2-7: Each subject's habitual food and fluid intake.
  Interventions: Other: Control

INTERVENTIONS:
Other: Water — Please see the associated arm description
  Arms: Water
Other: Coffee — Please see the associated arm description
  Arms: Coffee
Other: Control — Please see the associated arm description
  Arms: Control

SUMMARY:
39 healthy subjects without medication (except oral contraceptives) aged 20-70 years are recruited via advertisements or through telephone contacts with individuals that had previously participated in population-based cohort studies in Malmö. All subjects are exposed to three different intervention procedures; water and coffee loads (acutely and chronically), or no change from usual fluid intake (as a time-control), respectively in randomized order. The daily intake of coffee or water will amount to 3 L of water and 1 L of coffee, respectively for one week each. The three interventions (water, coffee and control), are separated by three weeks of normal fluid intake as a wash-out period.

By testing if simple life style interventions, i.e., increased water or coffee intake, may affect vasopressin secretion, evaluated as copeptin, we will increase the knowledge as to whether such life style induced changes of copeptin may in turn lead to effects on glucose tolerance as well as on other cardiometabolic risk factors previously shown to be associated with high copeptin level. Thus, the study will lead to further understanding about vasopressin and copeptin release and how life style manipulation of the vasopressin system may influence glucose metabolism and other cardiometabolic risk factors in healthy individuals.

DETAILED DESCRIPTION:
Day 1: The initial examination consists of medical history, clinical examination including office blood pressure, and blood sampling (overnight fasting plasma copeptin (a marker of vasopressin), osmolality, insulin, glucagon, glucose, creatinine, hsCRP and OGTT), and start of 24-h urine collection and 24-h ambulatory blood pressure measurement.

Day 2: After completion of the 24-h urine collection and ABPM, in the fasting state in the morning, office blood pressure will be measured and blood sampling for plasma copeptin, osmolality insulin, glucagon, glucose, creatinine and hsCRP measurement will be performed. Then, during a maximum time period of 20 minutes, subjects will ingest either 1L of water or 4 dL of coffee, or just 10 ml of water (time control). To map the acute coffee or water effect on copeptin, the experiment proceeds with repeated blood sampling every 30 minutes for 4 hours after the first coffee or water intake. Day 1 then continues with the rest of the daily intake, i.e., 2 L of water or 6 dL of coffee in addition to normal food and fluid intakes.

Day 3 to 7: 3 L water per day or 1 L of coffee per day are ingested (or nothing, in the control intervention) in addition to each subject's own food and fluid intake. On days 4 and 6, blood sampling for electrolyte and urea measurement and osmolality will be carried out for reasons of safety and compliance check.

Day 8: Fasting in the morning, office blood pressure, blood sampling (copeptin, osmolality, insulin, glucagon, glucose, creatinine, hsCRP) will be performed and a 24-h urine collection and ABPM will be started.

Day 9: The final examination will consist of clinical examination including office blood pressure and blood sampling (overnight fasting plasma copeptin, osmolality, insulin, glucagon, glucose, creatinine, hsCRP and OGTT), and end of 24-h urine collection and ABPM.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects Age 20-70 years

Exclusion Criteria:

medication (except oral contraceptives) any type of acute illness any type of chronic illness

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
1 week result on plasma copeptin | 7 days
  Change ("∆-value") between plasma copeptin value (pmol/L) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.

SECONDARY OUTCOMES:
1 week result on plasma glucose | 7 days
  Change ("∆-value") between plasma glucose (mmol/L) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
1 week result on plasma insulin | 7 days
  Change ("∆-value") between plasma insulin (IE) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
1 week result on plasma glucagon | 7 days
  Change ("∆-value") between plasma glucagon (pmol/L) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
1 week result on plasma C-reactive protein | 7 days
  Change ("∆-value") between plasma C-reactive protein (mg/L) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
1 week result on plasma creatinine | 7 days
  Change ("∆-value") between plasma creatinine (umol/L) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
1 week result on plasma osmolality | 7 days
  Change ("∆-value") between plasma osmolality (mosm/kg H2O) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
1 week result on urine osmolality | 7 days
  Change ("∆-value") between urine osmolality (mosm/kg H2O) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
1 week result on blood pressure | 7 days
  Change ("∆-value") between blood pressure (mmHg) at end of control week and post-intervention values will be calculated.
  Significance of differences between each intervention and the time-control will be tested using paired t-test or Wilcoxon's paired rank test, depending on normality of distributions.
Acute 4-hour effect of intervention on copeptin | 4 hours
  To test the hypothesis that acute coffee or water load affects plasma copeptin levels (pmol/L), we will perform paired t-tests (or Wilcoxon's paired rank test in case of no normal distribution) between individual 0 min values (immediately before acute load) and repeated post load values taken each 30 min during 4 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical research unit, Internal medicine department, Skåne University Hospital in Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No